CLINICAL TRIAL: NCT03298945
Title: Comparative Effectiveness of Split-Dose Colonoscopy Bowel Preparation Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-346
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy; colorectal cancer; bowel preparation regimen; pragmatic trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Golytely

STUDY DESIGN:
Intervention Model Description: Parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Golytely (Active Comparator): 4-L split-dose Golytely bowel prep
  Interventions: Drug: Golytely
- Miralax-Gatorade prep (Experimental): 2-L split-dose Miralax-Gatorade bowel prep
  Interventions: Drug: Miralax-Gatorade Prep

INTERVENTIONS:
Drug: Miralax-Gatorade Prep — 2-L split-dose Miralax-Gatorade bowel prep for colonoscopy
  Arms: Miralax-Gatorade prep
Drug: Golytely — 4-L split dose Golytely is the current standard prep at the VA
  Arms: Golytely

SUMMARY:
From the patients' perspective, the most formidable part of the colonoscopy experience is the process of bowel cleansing. A poorly tolerated bowel preparation regimen often leads to incompletion of scheduled colonoscopies which in turn undermines the effectiveness of colonoscopy, increases cost, and decreases patient satisfaction. The current standard bowel preparation in the VA is of larger volume and less palatable than another commonly used bowel preparation regimen. The investigators propose to compare these two commonly used bowel preparations with respect to the overall completion rate of scheduled colonoscopies in a real-world VA practice setting. The results of the study can be immediately applied to maximize the effectiveness of colonoscopy and increase patient satisfaction in the VA.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans Health Care: by identifying a colonoscopy bowel preparation regimen which is the most effective in real-world VA practice and can be immediately implemented on a VA-wide scale, the proposed study will maximize the effectiveness of colonoscopy in reducing colorectal cancer (CRC) risk among Veterans, increase Veteran satisfaction, and reduce VA healthcare cost. Background: CRC is a leading cause of cancer-related death among Veterans. Colonoscopy can effectively reduce CRC incidence and mortality. However, non-adherence to screening colonoscopy substantially undermines this benefit. Existing evidence indicates that a disagreeable bowel preparation is a leading barrier to completing a colonoscopy from the patients' perspective. The taste and the volume of the bowel preparation determine patient tolerability and compliance to the preparation instructions, which in turn affects the incompletion (e.g., cancellation/no-show/reschedule) rate of scheduled colonoscopies as well as the effectiveness of the completed colonoscopies and patient satisfaction. The two most commonly used preparations currently in the US are the split-dose 4L polyethylene glycol (PEG) and the split-dose 2L MiraLAX/Gatorade preparations. While a high-volume regimen may in theory be more effective than a lower volume one, it may be associated with lower tolerability and adherence in real-world practice. Three small trials have compared these two preparations. However, data from these explanatory trials cannot inform policy decisions because they were conducted under artificial conditions, restricted among narrow patient populations, and most importantly not designed to capture the full impact of bowel preparation on the completion rate or effectiveness of colonoscopy. To address this critical knowledge gap, the investigators are proposing a pragmatic trial to determine the optimal split-dose bowel preparation in the general Veteran population. Objectives: to compare the real-world effectiveness of the two most commonly used split-dose colonoscopy bowel preparation regimens in the US (i.e., 4L PEG and 2L MiraLAX/Gatorade) with respect to the completion rate of scheduled colonoscopies, adenoma detection rate and secondarily preparation quality, cancellation/no-show rate and patient-oriented outcomes (e.g., willingness to repeat the preparation).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age, and
* being scheduled for outpatient elective screening, surveillance or diagnostic colonoscopies, and
* the provider ordering the colonoscopy giving permission to enroll the patient.

Exclusion Criteria:

* Patients who are <18 years
* undergoing inpatient colonoscopy
* those with contra-indications to receiving the standard 4L PEG-ELS colonoscopy bowel preparation (e.g., allergy to PEG) will be excluded
* Those with a preference for a specific bowel preparation will be excluded.

  * The investigators are excluding inpatient colonoscopies because they account for a very small fraction of the total colonoscopies performed.
  * Also, inpatient colonoscopies are often performed for urgent reasons such that rapid bowel preparation procedures are followed.
* In addition, because the objective of inpatient colonoscopy is often not to look for small polyps, the threshold for "adequate" bowel preparation quality might be different from that for outpatient procedures.
* In addition, for patients undergoing more than 1 colonoscopy during the study period, only their first colonoscopy will be included in the primary analysis.
* Patients who are undergoing a repeat colonoscopy for to a recent inadequate colonoscopy examination with poor bowel preparation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2239 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Xiao Yang, MD MSCE, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comparative Effectiveness of Split-Dose Colonoscopy Bowel Preparation Regimens: A Pragmatic Randomized Controlled Trial Yang, Yu-Xiao, Dawei Xie, Raphael Rivero, Michael W. Bond, Jibreel Damisa, Qiao Lu, Nabeel H. Khan Gastroenterology, 2024-05-18, Volume 166, Issue 5, Pages S-353-S-353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on referral from the primary care providers ordering colonoscopy at the Corporal Michael J. Crescenz Department of Veterans Affairs Medical Center. The first participant was enrolled on December 13, 2018, and the last participant was enrolled on January 27, 2023.
Pre-assignment Details: Of the 3869 patients assessed for eligibility, 2239 met the eligibility criteria and were randomized.
Period: Overall Study
Arm/Group | Golytely | Miralax-Gatorade Prep
Started | 1139 | 1100
Completed | 1139 | 1100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golytely | Miralax-Gatorade Prep | Total
Number analyzed (Participants) | 1139 | 1100 | 2239
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.7) | 62.6 (9.5) | 62.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 113 | 220
  Male | 1032 | 987 | 2019
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 48 | 84
  Not Hispanic or Latino | 1074 | 1020 | 2094
  Unknown or Not Reported | 29 | 32 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 18 | 28
  Native Hawaiian or Other Pacific Islander | 9 | 18 | 27
  Black or African American | 407 | 397 | 804
  White | 670 | 631 | 1301
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 43 | 36 | 79
Body mass index group [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 10 | 9 | 19
  18.5 to 24.9 kg/m^2 | 198 | 175 | 373
  25 to 29.9 kg/m^2 | 395 | 368 | 763
  30 or more kg/m^2 | 527 | 543 | 1070
  Missing | 9 | 5 | 14
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 347 | 339 | 686
  Former smoker | 455 | 430 | 885
  Current smoker | 327 | 306 | 633
  Missing | 10 | 25 | 35
Alcohol use disorder [Count of Participants; unit: Participants] | 108 | 116 | 224
Diabetes mellitus [Count of Participants; unit: Participants] | 334 | 329 | 663
Constipation or narcotic use [Count of Participants; unit: Participants] | 19 | 22 | 41
Mental health disorders [Count of Participants; unit: Participants] | 371 | 398 | 769
Colonoscopy indications [Count of Participants; unit: Participants]
  Screening | 481 | 508 | 989
  Surveillance | 487 | 440 | 927
  Diagnostic | 171 | 152 | 323

OUTCOME MEASURES:

1. Primary Outcome: Colonoscopy Completion Rate
Description: The completion rate of scheduled colonoscopy will be defined as the proportion of patients who show up for their scheduled colonoscopy and have endoscopist-rated "adequate" bowel preparation quality, among those scheduled for a colonoscopy.
Time Frame: This outcome is determined within 1 month after colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Golytely | Miralax-Gatorade Prep
Number analyzed (Participants) | 1139 | 1100
Participants | 591 | 600

2. Primary Outcome: Population Level Adenoma Detection Rate (ADR)
Description: the ADR is estimated as the proportion of patients with at least one adenoma detected among all patients scheduled for colonoscopy.
Time Frame: within 1 month of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Golytely | Miralax-Gatorade Prep
Number analyzed (Participants) | 1139 | 1100
Participants | 383 | 364

3. Secondary Outcome: Cancellation or No-show in Each Bowel Prep Arm
Description: The proportion of patients who cancel or no-show in each group.
Time Frame: within 1 month after colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Golytely | Miralax-Gatorade Prep
Number analyzed (Participants) | 1139 | 1100
Participants | 358 | 330

4. Secondary Outcome: Adequate Bowel Prep Quality
Description: this is a binary indictor based on endoscopist rating of excellent or good quality bowel preparation
Time Frame: within 1 month after the colonoscopy
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patients With Inadequate Bowel Preparation Who Are Recommended to Have Earlier-than-usual Follow-up Colonoscopy
Description: patients with inadequate bowel preparation who are recommended to have earlier-than-usual follow-up colonoscopy
Time Frame: within 1 month after colonoscopy
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Hyponatremia
Description: Hyponatremia
Time Frame: within 6 months after colonoscopy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Renal Failure
Description: renal failure documented in CPRS
Time Frame: within 6 months of colonoscopy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Golytely | Miralax-Gatorade Prep
All-Cause Mortality (participants affected / at risk) | 7/1139 | 4/1100
Serious Adverse Events (participants affected / at risk) | 6/1139 | 5/1100
Other Adverse Events (participants affected / at risk) | 0/1139 | 0/1100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golytely (N=1139) | Miralax-Gatorade Prep (N=1100)
Colorectal cancer diagnosed on colonoscopy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Hospitalization for mania and psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for lung surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for DKA (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03298945/Prot_SAP_000.pdf